CLINICAL TRIAL: NCT06237920
Title: A Phase 2 Trial in Stage II-IIIa Urothelial Cancer Randomizing Pre-operative Nivolumab With or Without Relatlimab
Brief Title: Stage II-IIIa Urothelial Cancer Randomizing Pre-operative Nivolumab With or Without Relatlimab
Acronym: TURANDORELA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23TRR
Record Dates: First submitted 2023-11-10; First posted 2024-02-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Urinary Bladder Diseases; Male Urogenital Diseases; Urinary Bladder Neoplasm; Antineoplastics Toxicity
Keywords: Nivolumab; Relatlimab
MeSH Terms: conditions — Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Urinary Bladder Diseases; Male Urogenital Diseases; Urinary Bladder Neoplasms | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab (Experimental): 1 cycle of intravenous nivolumab on day 1 and 1 cycle of intraveous nivolumab on day 29. Total administration frequency is twice.
  Interventions: Drug: Nivolumab
- Nivolumab and relatlimab (Experimental): 1 cycle of intravenous nivolumab and relatlimab on day 1 and 1 cycle of intraveous nivolumab and relatlimab on day 29. Total administration frequency is twice.
  Interventions: Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Induction with immune checkpoint blockade nivolumab on day 1. Nivolumab will also be administered on day 29. Response evaluation will be after the last cycle of checkpoint inhibition.
  Other Names: Opdivo
Drug: Relatlimab — Induction with immune checkpoint blockade nivolumab and relatlimab on day 1. Nivolumab and relatlimab will also be administered on day 29. Response evaluation will be after the last cycle of checkpoint inhibition.
  Other Names: BMS-986016
  Arms: Nivolumab and relatlimab

SUMMARY:
This is a non-blinded phase 2 trial in Stage II-IIIa urothelial cancer randomizing pre-operative nivolumab with or without relatlimab to assess whether bladder preservation after dual immunotherapy would be a viable treatment option for patients responding to treatment

DETAILED DESCRIPTION:
This is a phase 2 study in which ninety adult patients with cT2-4aN0 or cT1-4aN1urothelial bladder cancer will be included.

Included patients will be treated with two cycles of checkpoint inhibition with nivolumab or two cycles of nivolumab+relatlimab every 28 days.

Response of this induction therapy will be evaluated by cystoscopy, mpMRI and a CT scan.

The primary endpoint is efficacy, defined as pathological complete response (pCR) defined as pT0N0 or pTisN0 at cystectomy.

Secondary end-points consist of feasibility analysis, defined as percentage of patients completing cystectomy within 12 weeks of start of treatment. Other key secondary end points are drug safety and overall and event-free survival. Events consist of death by any cause; disease recurrence inside or outside the urinary tract and switching to other treatments.

The first evaluation after completion of both treatment cycles will be after six months. Further follow-up visits will take place at 12 and 24 months after completion of the treatment. During these visits, focused physical examination, cystoscopy and a CT chest-abdomen will be performed, combined with registration of treatment-related adverse events and a questionnaire for evaluating QoL, bladder function and long-term effects of immunotherapy on QoL.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age ≥ 18 years
* Resectable muscle-invasive UC of the bladder, defined as cT2-4aN0M0 OR cT1-4aN1M0. In cT1N1 patients, lymph node positivity would need to be cytologically or histologically confirmed.
* Surgical resection (cystectomy) is the advised locoregional treatment and is accepted by the subject after consultation with the urologist.
* Patients are either cisplatin ineligible or elect to not undergo cisplatin based neoadjuvant chemotherapy after a balanced discussion of risks and benefits with the treating physician. Cisplatin eligibility is determined based on the Galsky criteria
* World Health Organization (WHO) performance Status 0 or 1.
* Urothelial cancer is the dominant histology (>50%). Any component of small cell or adenocarcinoma is not allowed.
* Formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks from diagnostic TUR available.
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, GFR>30 ml/min, AST ≤ 1.5 x ULN, ALT ≤1.5 x ULN, Bilirubin ≤1.5 X ULN
* Negative pregnancy test (βHCG in blood or urine) within 2 weeks of Day 1 Cycle 1 for female patients of childbearing potential.
* Highly effective contraception for female subjects if the risk of conception exists. Female patients of childbearing potential must comply with contraception methods as requested by the study protocol (→ 8.2.1 Pregnancy, contraception and breastfeeding)

Exclusion Criteria:

* Subjects with active autoimmune disease in the past 2 years. Patients with diabetes mellitus, properly controlled hypothyroidism or hyperthyroidism, vitiligo, psoriasis or other mild skin disease can still be included.
* Documented history of severe autoimmune disease (e.g. inflammatory bowel disease, myasthenia gravis).
* Previous intravenous systemic therapy or radiotherapy for UC.
* Upper urinary tract disease, unless all disease is planned to be resected in the same surgery as for UBC. This includes non-muscle-invasive disease.
* Prior CTLA-4, LAG3 or PD-1/PD-L1-targeting immunotherapy.
* Known active Human Immunodeficiency Virus infection, or tuberculosis, or other active infection:
* HIV-positive patients are eligible if the following applies:
* No AIDS defining opportunistic infection within the last year and a current CD4 count >350 cells/uL.
* Received antiretroviral therapy (ART) for at least 4 weeks prior to treatment and continued while enrolled on study
* CD4 counts and viral load are monitored per standard of care by a local health care provider
* In patients with a known history of hepatitis B or hepatitis C infection, Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA) should be negative
* Underlying medical conditions that, in the investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of adverse events. Examples may include severe pulmonary disease with extensive radiological abnormalities or intestinal disease causing severe diarrhea, not covered by other eligibility criteria, that may obscure colitis.
* Medical condition requiring the use of immunosuppressive medications, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) will be allowed.
* Use of other investigational drugs before study drug administration.
* Malignancy, other than urothelial cancer, in the previous 2 years, with a high chance of recurrence (estimated >10%). Patients with low-risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
* Pregnant and lactating female patients.
* Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
* Severe infections within 2 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, unstable arrhythmias and unstable angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | Immediately after surgery
  Pathological complete response defined as pT0N0 or pTisN0 in all evaluable patients

SECONDARY OUTCOMES:
Drug toxicity | Immunotherapy-related adverse events will be noted from time of immunotherapy start at day 1 throughout the study, up to 24 weeks after surgery.
  Safety in terms of immunotherapy-related adverse events according to CTCAE 5.0 criteria
Feasibility of dual immunotherapy | [Time Frame: From initiation of study drug until surgery, which will take place between day 50-71 after initiation of study drug]
  Percentage of patients that completes cystectomy within 12 weeks of start of treatment. Patients who elect to not undergo surgery or have a delay due to logistical reasons not related to study treatment will be excluded from this analysis.
Tumor tissue biomarkers predicting treatment response | 12 weeks after immunotherapy administration
  PD-L1 expression of tumor tissue (obtained pre-treatment) will be determined using immunohistochemistry of tissue slides. For PD-L1, tumor proportion score (TPS) will be determined. Pathological complete response will be related to PD-L1 expression
Exploring the Immunological effects of immunotherapy on the tumor microenvironment | 21 weeks after the last patient has started treatment
  RNA sequencing and multiplex immunofluorescence will be carried out on TUR and cystectomy tumor tissue. Methods may include RNA expression profiling and multiplex immunofluorescence.
Event-free survival | Through study completion, an average of 2 years
  Event-free survival is a composite endpoint, defined by the time from randomization to occurrence of any of the events below:
  * Disease recurrence outside the urinary tract (distant metastases, pelvic recurrence).
  * Disease progression precluding surgery.
  * Muscle invasive recurrence in the bladder or distal ureters in case surgery is not performed for other reasons than progression.
  * Switch to other treatments pre- or post-surgery directed at systemic UC (e.g. platinum-based chemotherapy combinations, antibody-drug conjugates etc.). In case adjuvant chemotherapy or immunotherapy is administered without evidence of residual disease, patients will be censored at the start of adjuvant therapy. Locoregional therapy to the bladder, such as (chemo)radiotherapy will not be considered an event in the absence of progressive disease.
Overall survival | Through study completion, an average of 2 years
  OS is defined as the time between the date of enrollment and the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Van der Heijden, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (9):
- Netherlands (9):
  - Rijnstate, Arnhem, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - NKI-AVL, Amsterdam, North Holland
  - Amsterdam UMC (AUMC), Amsterdam, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - ISALA, Zwolle, Overijssel
  - Leiden University Medical Center (LUMC), Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, Zuid_Holland
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No